CLINICAL TRIAL: NCT02637583
Title: Sequential Versus Simultaneous Vaccination With Pneumococcal Conjugate Vaccine (Prevenar 13) and Pneumococcal Polysaccharide Vaccine (Pneumovax 23) in Elderly: Immunological Memory and Antibody Levels
Brief Title: Sequential Versus Simultaneous Pneumococcal Vaccination in Elderly: Immunological Memory and Antibody Levels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Mathias Pletz, Prof. Dr. Mathias Pletz, Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EudraCT 2014-004013-85
Record Dates: First submitted 2015-10-21; First posted 2015-12-22 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Pneumococcal Infections
Keywords: conjugate vaccine; polysaccharide vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sequential vaccination PCV13 and PPV23 (Active Comparator): PCV13 0.5 ml intramuscular injection once on day 0 PPV23 0.5 ml intramuscular injection once 6 months later
  Interventions: Drug: PCV13; Drug: PPV23
- Simultaneous vaccination PCV13 and PPV23 (Experimental): PCV13 0.5ml intramuscular injection once on day 0 followed by PPV23 0.5ml intramuscular injection on day 0
  Interventions: Drug: PCV13; Drug: PPV23
- Single vaccinationPPV23 (Active Comparator): PPV23 0.5ml intramuscular injection on day 0
  Interventions: Drug: PPV23

INTERVENTIONS:
Drug: PCV13 — Intramuscular injection of 13-valent pneumococcal conjugate vaccine once
  Other Names: Prevenar 13
  Arms: Sequential vaccination PCV13 and PPV23; Simultaneous vaccination PCV13 and PPV23
Drug: PPV23 — Intramuscular injection of 23-valent pneumococcal polysaccharide vaccine once
  Other Names: Pneumovax (MSD)

SUMMARY:
The purpose of the present study is to compare the immunological response of pneumococcal serotype specific B-cells, the humoral immune response and safety after sequential vaccination versus simultaneous vaccination with 13-valent pneumococcal conjugate vaccine (PCV13) and 23-valent polysaccharide vaccine (PPV23) versus single vaccination with PPV23 in a prospective, randomized controlled monocentric head-to head clinical study in elderly. The hypothesis of this study is that simultaneous vaccination with PCV13 and PPV23 might achieve an improved immune-response compared to sequential vaccination or single vaccination.

Adults >=60 years without previous pneumococcal vaccination will be randomized in three groups and receive either PCV13 on day 0 plus PPV23 6 months later (sequential vaccination) or they receive PCV13 plus PPV23 simultaneous on day 0 (simultaneous vaccination) or they receive PPV23 on day 0 (single vaccination). Blood will be taken for pneumococcal serotype-specific B-memory cells against four vaccine-serotypes (ST), included in PCV13 and PPV23, vaccine-serotype 3 (ST3), vaccine-serotype 14 (ST14), vaccine-serotype 19A (ST19A) and vaccine-serotype 23F (ST23F) at visit 1, 2,4,5,7 and 8 and for antibody levels against the 12 vaccine-serotypes included in PCV13 and PPV23 at visit 1, 3, 4, 6, 7 and 8 in all three groups. Adverse events will be recorded for 28 days after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Unvaccinated adults >= 60 years
* Written informed consent

Exclusion Criteria:

* Hypersensitivity against substances included in both vaccines
* Previous pneumococcal vaccination
* Pneumonia within the last two months
* Active infection
* Autoimmune disease
* Ongoing or planned immunosuppressive therapy (including corticosteroid treatment with prednisolon equivalent dose >= 5 mg/d)
* Active malignant disease
* Drug abuse or alcoholic abuse
* Expectation of life < 2 years
* Coagulation disorders
* Burns or injury on the injection site
* Plegia or paresis of extremity where injection is planned
* Shock
* parallel participation in other clinical trial with intervention
* Infusion of blood products within the last half year

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Immune response of B-memory cells | 27-28 weeks after first vaccination
  Change of immune response of B memory cells against 4 pneumococcal serotypes ST3,ST14,ST19A und ST23F compared to day 0 will be determined by multiparameter flow cytometry. Pneumococcal specific B-cells will be identified by labeling with fluorochrome-coupled polysaccharide antigen, B-memory cells will be identified by expression of characteristic membrane proteins and quantified.

SECONDARY OUTCOMES:
Immune response of B-memory cells | 1-2 weeks, 26 weeks, 52 weeks, 104 weeks
  Change immune response of B memory cells against 4 pneumococcal serotypes ST3,ST14,ST19A und ST23F compared to day 0 will be determined by multiparameter flow cytometry. Pneumococcal specific B-cells will be identified by labeling with fluorochrome-coupled polysaccharide antigen, B-memory cells will be identified by expression of characteristic membrane proteins and quantified.
Humoral immune response | 4 weeks, 26 weeks, 30 weeks, 52 weeks, 104 weeks
  Change of serotype-specific immunoglobulin G concentrations against 12 pneumococcal vaccine-serotypes included in both vaccines PCV13 and PPV23 compared to day 0
Safety (Adverse events and serious adverse events) | 28 days after each vaccination
  Adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Pletz, MD, PhD, Principal Investigator — University Hospital of Jena, Center of Infectious Diseases and Infection Control
Locations (1):
- Center of Infectious Diseases and Infection Control, Jena University Hospital, Jena, Germany